CLINICAL TRIAL: NCT06857656
Title: Knowledge, Attitudes and Practices of Safe Handling of Cytotoxic Drugs Among Oncology Nurses and Clinical Pharmacists in Tertiary Care Unit
Brief Title: Knowledge, Attitudes and Practices of Safe Handling of CDs
Acronym: KAP CDs
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Younis Abdel Nazour, demonstrator at public health deprtment, Assiut University
Other Study IDs: KAP of handeling CDs
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Cytotoxic Drug
Keywords: occpational hazards

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cytotoic handular workers: Nurses and Clinical Pharmacists work in South Egypt Cancer Institute and Department of Clinical Oncology and Nuclear Medicine in Assiut university Hospital. At least one year of work experience in the hospital.
  Exposure to chemotherapy drugs

SUMMARY:
Cancer is a leading contributor to global disease burden, with nearly 20 million new cases diagnosed every year . Cancer patients usually receive a combination of treatments involving surgery, radiation, and/or systemic drug therapy.

Antineoplastic drugs (ADs), also known as chemotherapy or cytotoxic drugs, include compounds with various mechanisms of action that are used to fight the global burden of cancer, preventing or disrupting cell division of neoplastic cells. Also, Antineoplastic drugs are being used increasingly to treat arthritis, multiple sclerosis, and other non-cancer medical conditions.

However, their action on malignant cells is only partially selective and normal cells may also be affected, leading to significant toxic side effects.

Healthcare workers, particularly those working in oncology units, face the possibility of exposure to hazardous antineoplastic drugs, which are known to cause long-term health effects such as cancer, reproductive toxicity, and other chronic health issues. However, there is a gap in research specifically focused on exposure levels and health risks for nurses and pharmacists in tertiary care hospitals. Understanding the impact of this exposure and implementing proper preventive measures is crucial for ensuring the safety of healthcare workers.

The aim of the study:

General objectives: Evaluate the extent of exposure to a The widespread use of CDs has raised concern about the risks health care workers who use them.

Anyone working with patients (or animals) receiving cytotoxic drugs is at risk of exposure. This includes pharmacists, pharmacy technicians, medical and nursing staff, laboratory staff and Veterinary practitioners in which they are all at risk when using cytotoxics. Appropriate control measures must be in place to protect them all Occupational exposure to cytotoxic drugs (CDs) and related wastes may occur during preparing, administering, transporting, storing drugs and when handling cytotoxic waste, transporting and disposing of waste, and cleaning up spills. Exposure to those drugs may occur through skin absorption, inhalation of aerosols and drug droplets, eye contact through a splash of liquids, ingestion, and through needle stick injuries.

In Egypt, the burden of cancer is high; there is low number of nurses especially oncology certified nurses in compared to the patient's number. This makes nurses overwhelmed and frustrated, so, more exposed to CDs hazards.

Acute health effects related to this occupational exposure include hair loss, skin rash, eczema, skin flush, light headedness, nausea, dizziness, vomiting and gastrointestinal symptoms. While the long-term exposure may cause adverse reproductive outcomes including menstrual irregularities, infertility, spontaneous abortion and congenital malformation.

We need to mention results of previous studies Health care workers who handle CDs must be aware of the existing hazards and safe handling practices of cytotoxic drugs because this has been associated with improvement of safety of both patients and health care workers. Previous Egyptian studies show weak compliance of nurses' practice with safe-handling guidelines.

Safe handling of antineoplastic agents is a primary concern among health care workers (HCWs) due to the harmful effects of CDs. Various organizations like National Institute for Occupational Safety and Health (NIOSH), Occupational Safety and Health Administration (OSHA), American Society of Hospital Pharmacist (ASHP), the Oncology Nursing Society and American Society of Clinical Oncology (ASCO) have recommended safe handling practice guidelines for anti-cancer drugs. These guidelines suggest the application of hierarchy of various strategies of mitigating and controlling workplace hazards. All HCWs must follow these safety guidelines.

Some of the guidelines include modifying the physical structure of the workplace in terms of isolating the drug preparation space, minimizing nurses' contact with the drug, applying standard work methods and utilizing personal protective equipment to achieve the minimum contact of the antineoplastic drugs with the skin or respiratory system of HCWs.

A study was done in Ain Shams University Hospitals in 2019 by El Hosseini DM; Ghanem EA; Gamal DA and demonstrate that almost more than half of the study nurses frequently complained from recurrent headache (64.4%), skin irritation (63%), eye irritation (61.6%), and hair loss (52.1%). Reproductive effects were also found: menstrual irregularities (32.9%), low birth weight babies (23.3%), premature labor (19.2%), and malignancy (15.1%). During handling CDs, the majority of nurses (89%) utilized gloves, (61.6%) utilized gowns, and none of them utilized goggles. About (72. %) had fair total knowledge score regarding CDs, and only few of them (11.0 %) had good total In the last four decades, several studies have reported detectable and/or quantifiable concentrations of such hazardous drugs both in wor

DETAILED DESCRIPTION:
Cancer is a leading contributor to global disease burden, with nearly 20 million new cases diagnosed every year . Cancer patients usually receive a combination of treatments involving surgery, radiation, and/or systemic drug therapy.

Antineoplastic drugs (ADs), also known as chemotherapy or cytotoxic drugs, include compounds with various mechanisms of action that are used to fight the global burden of cancer, preventing or disrupting cell division of neoplastic cells. Also, Antineoplastic drugs are being used increasingly to treat arthritis, multiple sclerosis, and other non-cancer medical conditions.

However, their action on malignant cells is only partially selective and normal cells may also be affected, leading to significant toxic side effects.

Healthcare workers, particularly those working in oncology units, face the possibility of exposure to hazardous antineoplastic drugs, which are known to cause long-term health effects such as cancer, reproductive toxicity, and other chronic health issues. However, there is a gap in research specifically focused on exposure levels and health risks for nurses and pharmacists in tertiary care hospitals. Understanding the impact of this exposure and implementing proper preventive measures is crucial for ensuring the safety of healthcare workers.

The aim of the study:

General objectives: Evaluate the extent of exposure to a The widespread use of CDs has raised concern about the risks health care workers who use them.

Anyone working with patients (or animals) receiving cytotoxic drugs is at risk of exposure. This includes pharmacists, pharmacy technicians, medical and nursing staff, laboratory staff and Veterinary practitioners in which they are all at risk when using cytotoxics. Appropriate control measures must be in place to protect them all Occupational exposure to cytotoxic drugs (CDs) and related wastes may occur during preparing, administering, transporting, storing drugs and when handling cytotoxic waste, transporting and disposing of waste, and cleaning up spills. Exposure to those drugs may occur through skin absorption, inhalation of aerosols and drug droplets, eye contact through a splash of liquids, ingestion, and through needle stick injuries.

In Egypt, the burden of cancer is high; there is low number of nurses especially oncology certified nurses in compared to the patient's number. This makes nurses overwhelmed and frustrated, so, more exposed to CDs hazards.

Acute health effects related to this occupational exposure include hair loss, skin rash, eczema, skin flush, light headedness, nausea, dizziness, vomiting and gastrointestinal symptoms. While the long-term exposure may cause adverse reproductive outcomes including menstrual irregularities, infertility, spontaneous abortion and congenital malformation.

We need to mention results of previous studies Health care workers who handle CDs must be aware of the existing hazards and safe handling practices of cytotoxic drugs because this has been associated with improvement of safety of both patients and health care workers. Previous Egyptian studies show weak compliance of nurses' practice with safe-handling guidelines.

Safe handling of antineoplastic agents is a primary concern among health care workers (HCWs) due to the harmful effects of CDs. Various organizations like National Institute for Occupational Safety and Health (NIOSH), Occupational Safety and Health Administration (OSHA), American Society of Hospital Pharmacist (ASHP), the Oncology Nursing Society and American Society of Clinical Oncology (ASCO) have recommended safe handling practice guidelines for anti-cancer drugs. These guidelines suggest the application of hierarchy of various strategies of mitigating and controlling workplace hazards. All HCWs must follow these safety guidelines.

Some of the guidelines include modifying the physical structure of the workplace in terms of isolating the drug preparation space, minimizing nurses' contact with the drug, applying standard work methods and utilizing personal protective equipment to achieve the minimum contact of the antineoplastic drugs with the skin or respiratory system of HCWs.

A study was done in Ain Shams University Hospitals in 2019 by El Hosseini DM; Ghanem EA; Gamal DA and demonstrate that almost more than half of the study nurses frequently complained from recurrent headache (64.4%), skin irritation (63%), eye irritation (61.6%), and hair loss (52.1%). Reproductive effects were also found: menstrual irregularities (32.9%), low birth weight babies (23.3%), premature labor (19.2%), and malignancy (15.1%). During handling CDs, the majority of nurses (89%) utilized gloves, (61.6%) utilized gowns, and none of them utilized goggles. About (72. %) had fair total knowledge score regarding CDs, and only few of them (11.0 %) had good total In the last four decades, several studies have reported detectable and/or quantifiable concentrations of such hazardous drugs both in work

Rational of the study:

Healthcare workers, particularly those working in oncology units, face the possibility of exposure to hazardous antineoplastic drugs, which are known to cause long-term health effects such as cancer, reproductive toxicity, and other chronic health issues. However, there is a gap in research specifically focused on exposure levels and health risks for nurses and pharmacists in tertiary care hospitals. Understanding the impact of this exposure and implementing proper preventive measures is crucial for ensuring the safety of healthcare workers.

The aim of the study:

General objectives: Evaluate the extent of exposure to antineoplastic drugs among nurses and clinical pharmacists in a tertiary care unit and to examine the potential health effects associated with such exposure.

Specific objectives:

1. Determine the levels of exposure to antineoplastic drugs in the workplace among healthcare workers.
2. Compare the health status of those exposed to antineoplastic drugs with those who are not exposed.
3. Identify any protective measures that are currently in place and their effectiveness in reducing exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers (nurses and clinical pharmacists) employed in the tertiary care unit.

At least one year of work experience in the hospital. Exposure to chemotherapy drugs

Exclusion Criteria:

* Healthcare workers not involved in direct patient care or medication administration.

Workers with pre-existing conditions that may be influenced by factors unrelated to drug exposure (e.g., other environmental toxins).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthcare workers (nurses and clinical pharmacists) employed in the tertiary care unit.
  At least one year of work experience in the hospital. Exposure to chemotherapy drugs
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Total KAP score | baseline
  The knowledge score ranged from 0 to 26. Nurses who achieved ≥ 75% of the score (i.e. ≥ 20) were classified as having satisfactory knowledge, those who scored <75%were considered to have unsatisfactory knowledge. Regarding the attitude, the score ranged from 0 to 16. Nurses who achieved ≥ 75% of the attitude score (i.e. ≥ 12) were considered to have a positive attitude, while score less than 75% was considered as a negative one. For practice, the score ranged from 0 to 12. Nurses who obtained ≥ 75% of the score (i.e. ≥ 9) were classified as having adequate practice while those who achieved less than < 75% were classified as having inadequate practice. Total KAP ranged from 0-54, nurses who achieved ≥ 75% of the total score (≥ 41) were classified as having a satisfactory KAP, while obtaining less than 75% was considered as an unsatisfactory KAP.